CLINICAL TRIAL: NCT03098901
Title: Tc99m-PYP Scintigraphy in Order to Establish Incidence of Cardiac Transthyretin Amyloidosis Among Patients With Otherwise Unexplained Cardiomyopathies
Brief Title: Radioisotope Scintigraphy to Establish Incidence of Cardiac Amyloidosis Among Patients With Otherwise Unexplained Cardiac Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Sara Shimoni, Dr Sara Shimoni, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KMC-0018-17
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Cardiac TTR Amyloidosis
Keywords: TTR Amyloidosis; Heart Failure with Preserved Ejection Fraction; Ventricular arrhythmia; Cardiac Conduction Disturbances

STUDY DESIGN:
Intervention Model Description: Patients that suffer of one of the following conditions will be included in the study
  1. Patients suffering of HFpEF not explained by either hypertension or any other clinical condition.
  2. Patients with systolic dysfunction and non-significant coronary artery disease.
  3. Patients with diabetic cardiomyopathy
  4. Patients with otherwise unexplained left ventricular hypertrophy (LVH).
  5. Patients under age of 65 with idiopathic ventricular fibrillation (VF) or multiple ventricular premature beats (VPB) or ventricular tachycardia (VT) with a structurally normal heart.
  6. Patients under age of 65, with unexplained sinus node disease, sinoatrial block, complete or high-degree atrio-ventricular block or significant intraventricular conduction defect, with structurally normal heart whether having or not having received permanent implanted pacemaker.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- no other arm (Other)
  Interventions: Diagnostic Test: Tc99m-labeled pyrophosphate scan

INTERVENTIONS:
Diagnostic Test: Tc99m-labeled pyrophosphate scan — Intravenous injection of Tc99m-labeled pyrophosphate with consecutive whole body scan using gamma ray scanner for assessment of radioactive uptake in the heart. The results of the scan will be evaluated by a specialist in the field. The uptake will be graded using Perugini scale (0- no uptake, 1- uptake in heart less intense than in bones, 2-uptake in heart as intense as in bones, 3-uptake in heart more intense than in bones).

SUMMARY:
Cardiac amyloidosis is a multi-organ syndrome, which usually presents as restrictive cardiomyopathy (RCM). Transthyretin (TTR) amyloidosis (or ATTR) is a subtype of amyloidosis which frequently involves heart. Cardiac ATTR, though infrequently diagnosed during lifetime, may represent a prevalent cause of RCM, especially in elderly. Several medications that can limit progression of the disease are currently under investigation. Presently the golden standard for diagnosis of ATTR is endomyocardial biopsy (EMB) which may entail severe adverse complications causing under-diagnosis of ATTR.

Several papers support the evidence that Tc99m-labeled tracers can be used to detect myocardial deposits of TTR amyloid. It was suggested that Tc99m scintigraphy might be a highly sensitive diagnostic tool for cardiac ATTR. In this study the patients with otherwise unexplained cardiomyopathy or heart block will undergo Tc99m scan, which will establish the incidence of this largely underdiagnosed condition in the population.

DETAILED DESCRIPTION:
Amyloidosis is a multi-organ syndrome, which usually presents as a restrictive cardiomyopathy (RCM). Transthyretin (TTR) amyloidosis is a subtype of amyloidosis, further subdivided into familial type and senile type. Its pathophysiology consists primarily of abnormal precipitation of transthyretin - a protein that normally acts as transporter for thyroid hormone and retinoids - in tissues. TTR amyloidosis frequently involves heart, bringing about the same clinical and pathophysiological picture of RCM. Another presentation of TTR Amyloidosis can be atrio-ventricular block or bundle-branch block [1].

There is evidence that the cardiac TTR amyloidosis, though infrequently diagnosed during the lifetime, may represent a widespread cause of restrictive cardiomyopathy especially in elderly. An autopsy study in octogenarians having suffered of heart failure with preserved left ventricular ejection fraction (HFpEF) suggested that up to 25% of them had TTR amyloid deposit in myocardium, though a negligible minority of them had been diagnosed with TTR amyloidosis during their lifetime [2-3]. HFpEF is a very widespread diagnosis, which represents a considerable burden of morbidity, and usually harbours populations of patients poorly responding to treatment. Most of patients with the diagnosis of HFpEF have little or no explanation concerning the aetiology of their disease, especially if they do not respond to conventional treatment. Most of them can benefit only from symptomatic treatment which does not alter the course of the disease. Thus a more widespread diagnosis of TTR amyloidosis could have been very promising as to a better management of this hard-to-treat patient population.

Several medications that can limit progression of TTR amyloidosis are currently under investigation. Until now, the golden standard for diagnosis of the disease was endomyocardial biopsy (EMB) which may entail several adverse complications and thus limit widespread diagnosis. Since amyloidosis is a multi-organ disease, extra-cardiac biopsy was proposed as a surrogate tissue diagnosis, though in TTR amyloidosis its sensitivity is below 50% [4].

Recently several papers support the evidence that Tc99m-labeled pyrophosphate (PYP) and bisphosphonates when injected intravenously localize to myocardial deposits of TTR amyloid. It was thus suggested that Tc99m scintigraphy might be a highly sensitive and specific diagnostic tool for cardiac TTR amyloidosis [5-9]. It was shown that almost the only source of false positive Tc99m scintigraphy is primary amyloidosis, which is a different entity, with worse prognosis, different treatment, although frequently involves heart as well [10]. Primary amyloidosis can be diagnosed by means of demonstration of monoclonal immunoglobulin peak in serum and immunoglobulin light chains in serum and urine [11]. Therefore, the specificity of Tc99m scan for TTR amyloidosis can be brought to an extraordinary level, with virtually negligible false positive rate, if primary amyloidosis is excluded prior to referral to Tc99m scan. The other entity where false positive uptake of Tc99m in myocardium can be observed is acute myocardial infarction. Currently the Tc99m-PYP scan is utilised as bone scan according to guidelines in order to diagnose wide spectrum of diseases such as stress fractures or metastatic bone disease.

At present the mentioned hypothesis that TTR amyloidosis might be a widespread cause of HFpEF has not been established in a clinical trial due to the fact that until now the most accurate diagnosis of TTR amyloidosis required an invasive procedure with possible adverse outcomes while the extra-cardiac biopsy had low diagnostic yield. Advent of a novel, possibly as accurate, yet non-invasive diagnostic tool opens new opportunities to set such study.

The incidence of both familial type and senile type TTR amyloidosis among patients with diagnosis of otherwise unexplained heart failure or heart block will be evaluated in this study by means of Tc99m scan using SPECT technology as described above. The hypothesis is that if the incidence of TTR amyloidosis within the population of patients suffering of HFpEF is as high as it was demonstrated by the autopsy studies, then we will be able to establish the diagnosis in a larger cohort of patients. This will make new developments in the research of the disease, such as treatment and outcome driven trials, possible.

Establishing the diagnosis of TTR amyloidosis in patients with HFpEF will improve our decision-making ability regarding the patients' treatment, for example preventing unnecessary invasive measures in patients with comorbidities demanding such measures, the alternative diagnoses being unrevealed.

ELIGIBILITY:
Inclusion Criteria:

1. Heart Failure with Preserved Ejection Fraction not explained by either hypertension or any other clinical condition.
2. Systolic dysfunction and non-significant coronary artery disease.
3. Diabetic cardiomyopathy
4. Otherwise unexplained left ventricular hypertrophy (LVH).
5. Under age of 65 and idiopathic ventricular fibrillation (VF) or multiple ventricular premature beats (VPB) or ventricular tachycardia (VT) with a structurally normal heart.
6. Under age of 65, and unexplained sinus node disease, sinoatrial block, complete or high-degree atrio-ventricular block or significant intraventricular conduction defect, with structurally normal heart whether having or not having received permanent implanted pacemaker.

Exclusion Criteria:

1. Primary amyloidosis cannot be excluded,
2. Acute or recent (3 months) myocardial infarction,
3. Acute or recent (12 months) myocarditis,
4. Oncologic or any other co-morbidity, which can shorten the patient's survival to less than one year,
5. End stage renal disease treated with dialysis,
6. Ischemic cardiomyopathy,
7. Non-TTR amyloidosis known or suspected,
8. Another type of cardiomyopathy (for ex. arrhythmogenic right ventricular dysplasia),
9. Any disease or clinical condition that can lead to cardiomyopathy (history of anthracyclines treatment, history of alcohol abuse, multiple myeloma, sarcoidosis, carcinoid, inflammatory and autoimmune diseases).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-15 (Estimated); Primary Completion 2018-04-15 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
diagnosis or exclusion of any type of cardiac amyloidosis; | immediately at the Tc99m scan performing or within a year form beginning of the recruitment
  diagnosis of cardiac TTR amyloidosis, or any other type of cardiac amyloidosis, or diagnosis of another condition other than amyloidosis explaining the patient's clinical cardiological findings

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruberg FL, Berk JL. Transthyretin (TTR) cardiac amyloidosis. Circulation. 2012 Sep 4;126(10):1286-300. doi: 10.1161/CIRCULATIONAHA.111.078915. No abstract available. PMID 22949539
- [Background] Tanskanen M, Peuralinna T, Polvikoski T, Notkola IL, Sulkava R, Hardy J, Singleton A, Kiuru-Enari S, Paetau A, Tienari PJ, Myllykangas L. Senile systemic amyloidosis affects 25% of the very aged and associates with genetic variation in alpha2-macroglobulin and tau: a population-based autopsy study. Ann Med. 2008;40(3):232-9. doi: 10.1080/07853890701842988. PMID 18382889
- [Background] Fine NM, Arruda-Olson AM, Dispenzieri A, Zeldenrust SR, Gertz MA, Kyle RA, Swiecicki PL, Scott CG, Grogan M. Yield of noncardiac biopsy for the diagnosis of transthyretin cardiac amyloidosis. Am J Cardiol. 2014 May 15;113(10):1723-7. doi: 10.1016/j.amjcard.2014.02.030. Epub 2014 Mar 2. PMID 24698461
- [Background] Maurer MS. Noninvasive Identification of ATTRwt Cardiac Amyloid: The Re-emergence of Nuclear Cardiology. Am J Med. 2015 Dec;128(12):1275-80. doi: 10.1016/j.amjmed.2015.05.039. Epub 2015 Jun 17. PMID 26091765
- [Background] Perugini E, Guidalotti PL, Salvi F, Cooke RM, Pettinato C, Riva L, Leone O, Farsad M, Ciliberti P, Bacchi-Reggiani L, Fallani F, Branzi A, Rapezzi C. Noninvasive etiologic diagnosis of cardiac amyloidosis using 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy. J Am Coll Cardiol. 2005 Sep 20;46(6):1076-84. doi: 10.1016/j.jacc.2005.05.073. PMID 16168294
- [Background] Rapezzi C, Quarta CC, Guidalotti PL, Longhi S, Pettinato C, Leone O, Ferlini A, Salvi F, Gallo P, Gagliardi C, Branzi A. Usefulness and limitations of 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy in the aetiological diagnosis of amyloidotic cardiomyopathy. Eur J Nucl Med Mol Imaging. 2011 Mar;38(3):470-8. doi: 10.1007/s00259-010-1642-7. Epub 2010 Nov 11. PMID 21069320
- [Background] Bokhari S, Castano A, Pozniakoff T, Deslisle S, Latif F, Maurer MS. (99m)Tc-pyrophosphate scintigraphy for differentiating light-chain cardiac amyloidosis from the transthyretin-related familial and senile cardiac amyloidoses. Circ Cardiovasc Imaging. 2013 Mar 1;6(2):195-201. doi: 10.1161/CIRCIMAGING.112.000132. Epub 2013 Feb 11. PMID 23400849
- [Background] Gillmore JD, Maurer MS, Falk RH, Merlini G, Damy T, Dispenzieri A, Wechalekar AD, Berk JL, Quarta CC, Grogan M, Lachmann HJ, Bokhari S, Castano A, Dorbala S, Johnson GB, Glaudemans AW, Rezk T, Fontana M, Palladini G, Milani P, Guidalotti PL, Flatman K, Lane T, Vonberg FW, Whelan CJ, Moon JC, Ruberg FL, Miller EJ, Hutt DF, Hazenberg BP, Rapezzi C, Hawkins PN. Nonbiopsy Diagnosis of Cardiac Transthyretin Amyloidosis. Circulation. 2016 Jun 14;133(24):2404-12. doi: 10.1161/CIRCULATIONAHA.116.021612. Epub 2016 Apr 22. PMID 27143678
- [Background] Kyle RA, Gertz MA. Primary systemic amyloidosis: clinical and laboratory features in 474 cases. Semin Hematol. 1995 Jan;32(1):45-59. No abstract available. PMID 7878478